CLINICAL TRIAL: NCT00005768
Title: Estrogen Modulation of Mood and Cognition Following Monoaminergic Depletion in Post-Menopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00109-0741; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Menopause
MeSH Terms: interventions — Estrogens

INTERVENTIONS:
Drug: Estrogen

SUMMARY:
This study will examine whether estrogen administration in postmenopausal women can alter the response to changes in brain chemistry brought about by dietary manipulation. Women who are recently menopausal (50-60 yrs. of age) and over 20 years postmenopausal (>70 yrs. of age) will take estrogen or placebo for three months. At the end of that time they will participate in three challenges using dietary techniques to briefly change the relative amounts of neurotransmitters in the brain that are believed to be related to mood regulation (serotonin, dopamine, and norepinephrine). Previous research has shown that these dietary manipulations can briefly produce negative changes in mood. The investigator hypothesizes that estrogen administration will blunt or buffer these negative effects in a quantifiable way. The investigator believes that this will provide a direct test of the ability of estrogen to meaningfully change the brain chemistry of mood in a clinically measurable and positive way. The proposed procedure will also allow assessment of the effects of estrogen on brain neurotransmitter systems after many years of very low estrogen levels.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Non-smoker
* BMI <30
* Healthy
* Without surgically-induced menopause
* Not on HRT or >1 year post HRT
* Normal mammogram within last year
* No cardiovascular disease other than mild hypertension

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States